CLINICAL TRIAL: NCT03504800
Title: Optical Coherence Tomography-Aided Differential Diagnosis and Treatment of Irregular Corneas
Brief Title: OCT in Diagnosis of Irregular Corneas
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Yan Li, PhD, Assistant Professor of Ophthalmology, Oregon Health and Science University
Other Study IDs: IRB#000018036
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus; Corneal Opacity; Corneal Dystrophy
Keywords: OCT; Keratoconus
MeSH Terms: conditions — Keratoconus; Corneal Opacity; Corneal Dystrophies, Hereditary | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group A: Classification of Corneal Irregularities: This group will consist of participants >14 years old with various types of corneal irregularities. Their data will be compared against participants with healthy corneas. Data for this group will be gathered only once.
  Interventions: Device: Optical Coherence Tomography
- Group B: Detection of Keratoconus Progression: Participants from Group A who are diagnosed with keratoconus will be selected for this longitudinal study to monitor keratoconus progression. They will be followed up to 4 years.
  Interventions: Device: Optical Coherence Tomography
- Group C: OCT-and-Topography Guided PTK: Participants from Group A will be selected for this group if they have vision primarily limited by scars, dystrophy, or high astigmatism that could be treated by PTK. They will be followed up to 1 year.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — This device will be used to tightly classify corneal irregularities and determine eligibility of candidates from Group A into Groups B & C.

SUMMARY:
This main goal of this study is to improve the detection, classification, monitoring, and treatment of irregular corneas due to keratoconus, warpage, dry eye, scar, stromal dystrophies, and other corneal conditions.

The primary goal will be achieved by using optical coherence tomography (OCT) to:

1. Develop an OCT-based system to classify and evaluate corneal-shape irregularities.
2. Develop OCT metrics for more sensitive detection of keratoconus progression.
3. Develop OCT-and-topography guided phototherapeutic keratectomy (PTK) for irregular corneas.

ELIGIBILITY:
Inclusion Criteria:

GROUP A:

* Keratoconus:

  1. CDVA ≥ 20/25 in the better eye; and both of the following in the worse eye
  2. Topography characteristic of keratoconus or pellucid marginal degeneration
* Contact lens-related corneal warpage:

  1. Contact lens use; and
  2. Topography irregularities
* Dry eye:

  1. Symptoms of dry eye documented by Ocular Surface Disease Index (OSDI) questionnaire score ≥ 30; and
  2. Topography irregularities
  3. Presence of punctate epithelial erosion on exam with surface staining
  4. Aqueous deficiency or evaporative dry eye
* Epithelial basement membrane dystrophy (EBMD):

  1. Negative corneal fluorescein staining; and
  2. Corneal opacities; and
  3. Topography irregularities
* Stromal addition or subtraction:

  1. Scars; or
  2. Salzmann's degeneration; or
  3. Stromal dystrophies; or
  4. Complication (visual complaints) after LASIK or photorefractive keratectomy (PRK)
* Stromal distortion:

  1. Radial keratectomy (RK); or
  2. Corneal transplants.
* Normal controls:

  1. Healthy eyes with no previous eye procedures/surgeries.

GROUP B:

Participants will be selected from the keratoconus population in Group A based on topography findings.

GROUP C:

Participants will be selected from the stromal addition/subtraction and stromal distortion populations of Group A if they have vision primarily limited by scars, dystrophy, or high astigmatism that could benefit from PTK.

Exclusion Criteria (all groups):

* Inability to give informed consent.
* Inability to maintain fixation for OCT imaging.
* Inability to commit to required study visits.
* Eyes with concurrent cataract, retinal disease, glaucoma, or other eye conditions that may limit the visual outcome after surgery.
* Previous corneal surgeries if considered as a keratoconus participant.
* Pregnancy or breastfeeding.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 445 participants ages 14 or older will be recruited for the 3 clinical studies. All 3 studies will be performed at the Casey Eye Institute at Oregon Health & Science University.
  Group A:
  * Keratoconus: 150 participants
  * Epithelial deformation: 105 participants; This category includes contact lens-related corneal warpage, dry eye, and EBMD.
  * Primary stromal changes: 100 participants; This category includes corneal scars, Salzmann's degeneration, stromal dystrophies, complicated LASIK/PRK cases with visual complaints, RK cases, and corneal transplants.
  * Healthy Controls: 90 participants
Sampling Method: Non-Probability Sample
Enrollment: 445 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Develop OCT-based system to classify and evaluate corneal-shape irregularities | 1 day
  Clinical classification of keratoconus, epithelial deformation, stromal addition/subtraction, stromal distortion, and healthy controls by OCT. Primary measurements will be corneal and epithelial thicknesses assessed in micron units.
Develop OCT-based system to classify and evaluate corneal-shape irregularities | 1 day
  Secondary measurement will be OCT corneal shape assessed in Diopter units.
Develop OCT metrics for more sensitive detection of keratoconus progression | 4 year
  Primary measurements will be OCT corneal and epithelial thicknesses assessed in micron units.
Develop OCT metrics for more sensitive detection of keratoconus progression | 4 year
  Secondary measurement will be OCT corneal shape assessed in Diopter units.
Develop OCT- and topography-guided phototherapeutic keratectomy (PTK) for irregular corneas | 1 year
  The primary goal is to improve the post-procedural outcome of uncorrected and best corrected visual acuity. This will be measured in feet by conventional Snellen fraction of 20/xx.
Develop OCT- and topography-guided phototherapeutic keratectomy (PTK) for irregular corneas | 1 year
  The secondary goal is to improve the post-procedural outcome of refractive error. This will be measured in Diopter units.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Humberto Martinez, Portland, Oregon, United States